CLINICAL TRIAL: NCT01006278
Title: Molecular Biomarkers Associated With Degenerative Joint Disease
Brief Title: Molecular Biomarkers Associated With Degenerative Joint Disease in the Knee
Status: Completed | Type: Observational
Sponsor: Scuderi, Gaetano J., M.D. (Other)
Collaborators: Stanford University (Other)
Responsible Party: Gaetano J Scuderi, MD, Stanford University
Other Study IDs: Cyt.002
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Cartilage Diseases
Keywords: biomarker; knee arthroscopy; pain
MeSH Terms: conditions — Cartilage Diseases; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — synovial fluid ananysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgical group with knee pain: patients 18 years of age or greater with a history of knee pain for more than three but less than six months who failed conservative management with the presence of mechanical symptoms including locking, catching, or giving way; positive physical exam findings including joint line tenderness, McMurray's exam, or Steinman's exam; and MRI of the knee positive for meniscus tear in a location correlating with physical examination. Exclusion criteria were as follows: the presence of high grade gonarthrosis including Kellgren-Lawrence grade IV; a history of prior knee surgery or trauma; ligamentous incompetence on examination or MRI; and diagnosis of inflammatory arthritides, crystalline arthropathies, or other rheumatologic diseases.
- Group 2: volunteer group

SUMMARY:
This investigation describes a novel complex of structural degradation proteins that is associated with pain in individuals with meniscal pathology undergoing arthroscopic partial meniscectomy. The presence of the complex in the synovial fluid of the knee is sensitive and specific for the painful state compared with similar aged controls. The absence of the complex in asymptomatic controls makes it a useful biomarker for the disease state.

DETAILED DESCRIPTION:
Background: Molecular biomarkers associated with knee pain may be useful as diagnostic tools, prognostic indicators, and surrogate endpoints for therapeutic trials. This study describes a novel complex of structural degradation proteins which are present in the knees of patients with meniscal pathology.

Methods: This prospective cohort study included 30 patients with knee pain, mechanical symptoms, and MRI positive for meniscus tear who elected for arthroscopic partial meniscectomy after failing conservative management. Synovial fluid was aspirated at the time of surgery and assayed for a complex of structural degradation proteins by means of heterogeneous ELISA. The results were compared to knee aspirates from 10 asymptomatic volunteers with no pain. The complex was identified by a proteomic analysis of including multiplexed-bead immunoassay, purification by anion exchange and size exclusion chromatography, and mass spectrometry of individual chromatographic fractions.

ELIGIBILITY:
Inclusion Criteria:

* the presence of mechanical symptoms including locking, catching, or giving way;
* positive physical exam findings including joint line tenderness, McMurray's exam, or Steinman's exam; and
* MRI of the knee positive for meniscus tear in a location correlating with physical examination.

Exclusion Criteria:

* the presence of high grade gonarthrosis including Kellgren-Lawrence grade IV;
* a history of prior knee surgery or trauma; ligamentous incompetence on examination or MRI; and
* diagnosis of inflammatory arthritides, crystalline arthropathies, or other rheumatologic diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The operative group consisted of patients 18 years of age or greater with a history of knee pain for more than three but less than six months who failed conservative management including NSAIDs, physical therapy, and activity modification.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano J Scuderi, MD, Principal Investigator — Stanford University